CLINICAL TRIAL: NCT04517305
Title: Pyrotinib Plus Vinorelbine in Metastatic HER2-positive Breast Cancer Patients- a Multicenter Retrospective Study
Brief Title: Pyrotinib Plus Vinorelbine in HER2+ Metastatic Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-10
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: Pyrotinib
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pyrotinib plus vinorelbine: Patients used pyrotinib plus vinorelbine as treatment for metastatic breast cancer.

SUMMARY:
To evaluate the patterns and treatment outcomes of pyrotinib plus vinorelbine in the real world.

ELIGIBILITY:
Inclusion Criteria:

* woman, age > 18 years old
* diagnosed with HER2 +Metastatic Breast Cancer
* pyrotinib plus vinorelbine for at least one cycle, starting from 2018.05-2020.05
* available medical history

Exclusion Criteria:

* medical history was incomplete

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to International Classification of Diseases-10, ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Y, Qiu Y, Li H, Luo T, Li W, Wang H, Shao B, Wang B, Ge R. Pyrotinib Combined With Vinorelbine in HER2-Positive Metastatic Breast Cancer: A Multicenter Retrospective Study. Front Oncol. 2021 Apr 20;11:664429. doi: 10.3389/fonc.2021.664429. eCollection 2021. PMID 33996589